CLINICAL TRIAL: NCT07101679
Title: A Phase II Clinical Study of GnP Regimen (Nab-paclitaxel + Gemcitabine) Combined With Serplulimab and Stereotactic Body Radiation Therapy (SBRT) as First-line Treatment for Locally Advanced Pancreatic Cancer
Brief Title: A Study of GnP RegimenCombined With Serplulimab and Stereotactic Body Radiation Therapy as First-line Treatment for Locally Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Dan Cao, professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025(247)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma
Keywords: SBRT; serplulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LICSBR GROUP (Experimental): Participating patients will receive the GnP regimen every 21 days (nab-paclitaxel 125mg/m² ivgtt on days 1 and 8 + gemcitabine 1000mg/m² ivgtt on days 1 and 8, repeated every 21 days) combined with serplulimab (200mg ivgtt Q3W). In the second cycle, patients will receive SBRT targeting the primary tumor and/or retroperitoneal lymph nodes: 6.6Gy×5 fractions, 7Gy×5 fractions, or 8Gy×5 fractions, administered every other day with radiotherapy completed in 5 sessions (specific selection determined by investigators based on lesion size and organs at risk [OAR] assessment). Comprehensive evaluation including tumor markers and CT scans will be performed every 2 cycles with multidisciplinary team (MDT) review, and patients who meet surgical criteria will undergo radical resection surgery.本研究为单臂 II 期临床试验。研究目标为年龄在 18-75 岁之间、ECOG 体能状态评分为 0-2 分、经病理学和影像学综合评估（CT 或 MRI）确诊为局部晚期胰腺导管腺癌的患者。参与患者将接受 GnP 方案治疗，每 21 天一次（第 1 天和第 8 天给予 nab-紫杉醇 125mg/m²静脉滴注，第 1 天和第 8 天给予吉西他滨 1000mg/m²静脉滴注，每 21 天重复一次），联合塞普卢利单抗（
  Interventions: Drug: LICSBR

INTERVENTIONS:
Drug: LICSBR — Participating patients will receive the GnP regimen every 21 days (nab-paclitaxel 125mg/m² ivgtt on days 1 and 8 + gemcitabine 1000mg/m² ivgtt on days 1 and 8, repeated every 21 days) combined with serplulimab (200mg ivgtt Q3W). In the second cycle, patients will receive SBRT targeting the primary tumor and/or retroperitoneal lymph nodes: 6.6Gy×5 fractions, 7Gy×5 fractions, or 8Gy×5 fractions, administered every other day with radiotherapy completed in 5 sessions (specific selection determined by investigators based on lesion size and organs at risk [OAR] assessment).

SUMMARY:
This study is a single-arm phase II clinical trial. The study targets patients aged 18-75 years with ECOG performance status 0-2, diagnosed with locally advanced pancreatic ductal adenocarcinoma based on comprehensive assessment of pathology and imaging studies (CT or MRI). Participating patients will receive the GnP regimen every 21 days (nab-paclitaxel 125mg/m² ivgtt on days 1 and 8 + gemcitabine 1000mg/m² ivgtt on days 1 and 8, repeated every 21 days) combined with serplulimab (200mg ivgtt Q3W). In the second cycle, patients will receive SBRT targeting the primary tumor and/or retroperitoneal lymph nodes: 6.6Gy×5 fractions, 7Gy×5 fractions, or 8Gy×5 fractions, administered every other day with radiotherapy completed in 5 sessions (specific selection determined by investigators based on lesion size and organs at risk [OAR] assessment). Comprehensive evaluation including tumor markers and CT scans will be performed every 2 cycles with multidisciplinary team (MDT) review, and patients who meet surgical criteria will undergo radical resection surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria (1)Histologically confirmed pancreatic ductal adenocarcinoma with diagnosis based on comprehensive assessment of pathology and imaging studies (CT or MRI), supplemented by fibroblast activation protein positron emission tomography-computed tomography (FAPI PET-CT) when necessary, determined as locally advanced pancreatic cancer by multidisciplinary team assessment (per 2022 CSCO guideline definition) and deemed unresectable; (2)Treatment-naïve patients with no prior anticancer therapy (including chemotherapy, radiotherapy, surgery, radiofrequency ablation, irreversible electroporation, or other investigational treatments); (3)Age 18-75 years, inclusive, regardless of sex; (4)Eastern Cooperative Oncology Group (ECOG) performance status 0-2; (5)Measurable primary tumor lesions: ≥10 mm in longest diameter on spiral CT, lymph nodes ≥15 mm in short axis diameter; for conventional CT or physical examination, maximum diameter must be ≥20 mm; (6)Adequate major organ function:

   * Bone marrow function (no blood transfusion within 14 days prior to screening): White blood cell count (WBC) ≥4.0×10⁹/L, absolute neutrophil count (ANC) ≥1.5×10⁹/L, platelet count (PLT) ≥80×10⁹/L, hemoglobin (Hb) ≥90 g/L;
   * Hepatic function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3× upper limit of normal (ULN), total bilirubin (TBIL) ≤2×ULN (for subjects with hepatic metastases: ALT and AST ≤5×ULN, TBIL ≤2×ULN), Child-Pugh score ≤7;
   * Renal function: Serum creatinine (Cr) ≤1.5×ULN, proteinuria ≤2+ or ≤2 g/24h, glomerular filtration rate (GFR) ≥60 mL/min/1.73 m²;
   * Coagulation function: Prothrombin time (PT), activated partial thromboplastin time (aPTT), and international normalized ratio (INR) ≤1.5×ULN. Patients receiving stable anticoagulation therapy for at least 30 days prior to study drug treatment may have PT or INR >1.5×ULN if deemed appropriate for the study by investigator assessment, provided adequate justification is documented;
   * Serum sodium, potassium, calcium, and magnesium levels ≤Grade 1 per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0;
   * Electrocardiogram showing corrected QT interval (QTc) ≤480 ms; (7)No history of autoimmune disease or current autoimmune disease; (8)Life expectancy ≥3 months; (9)Signed written informed consent prior to any study-related procedures, with ability to understand the protocol and comply with study requirements.

Exclusion Criteria:

1. Known hypersensitivity or allergy to any of the study drugs;
2. Patients with distant metastatic disease classified as Stage IV pancreatic cancer;
3. Patients whose tumor lesions are determined by the surgical team or multidisciplinary team to be resectable or borderline resectable pancreatic cancer based on imaging studies (CT or MRI) (per 2022 CSCO guideline definition);
4. Patients whose lesions are deemed unsuitable for stereotactic body radiation therapy (SBRT) by investigator assessment;
5. Known or suspected central nervous system (CNS) metastases, defined as subjects with signs or symptoms suggestive of CNS metastases, unless CNS metastases have been excluded by CT or MRI;
6. History of other malignancies within 5 years (except adequately treated basal cell carcinoma of the skin and cervical carcinoma in situ);
7. Requirement for concurrent anticancer treatments other than the study treatment regimen during the study period, including chemotherapy, targeted therapy, hormonal therapy, immunotherapy regimens, radiotherapy, or traditional Chinese medicine with anticancer properties;
8. Prior or current use of chemotherapy, focal adhesion kinase (FAK) inhibitors, or anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibodies (including ipilimumab or any other antibody or drug targeting T-cell co-stimulation or checkpoint pathways);
9. Diagnosis of immunodeficiency or receiving chronic systemic corticosteroid therapy (daily dose exceeding 10 mg prednisone or equivalent) or any other form of immunosuppressive treatment within 7 days prior to first study drug administration;
10. Receipt of live vaccines within 30 days prior to first study drug treatment (including but not limited to: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, bacillus Calmette-Guérin [BCG], and typhoid vaccines). Inactivated vaccines such as injectable seasonal influenza vaccines are permitted, but live attenuated vaccines such as intranasal influenza vaccines (e.g., FluMist) are not allowed;
11. Uncontrolled hypertension (defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg despite treatment);
12. Significant cardiac disease, including congestive heart failure (New York Heart Association [NYHA] Class III-IV), prior myocardial infarction, or uncontrolled angina within 6 months;
13. Cardiac arrhythmias requiring treatment, including atrial fibrillation, supraventricular tachycardia, ventricular tachycardia, or ventricular fibrillation; confirmed ECG abnormalities deemed by the investigator to require clinical intervention or treatment;
14. History of hemorrhagic or thromboembolic events within 6 months, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, or spontaneous major tumor bleeding;
15. Need for surgical treatment within 28 days before or anticipated within 28 days after the last study drug administration;
16. Presence of poorly controlled third-space fluid collections, such as large pleural effusions or ascites;
17. istory of gastrointestinal perforation or suspected risk of gastrointestinal perforation;
18. Investigator determination that concomitant medications required during the study period may affect study drug metabolism, such as strong CYP3A4 inhibitors or inducers, drugs primarily metabolized by CYP3A4, 2C8, 2C9, 2C19, or 2D6 with narrow therapeutic indices;
19. Severe psychiatric disorders;
20. Pregnancy, potential pregnancy, or lactation;
21. Subjects of childbearing potential unwilling to use contraception during the study period and for 3 months after the last study drug administration;
22. Participation in other drug or medical device clinical trials within 4 weeks prior to study entry;
23. Any condition deemed inappropriate for study participation by investigator judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed Objective Response Rate (ORR) | 4 YEARS
  The proportion of subjects in the intention-to-treat (ITT) population who achieve a best overall response of complete response (CR) or partial response (PR) during the study treatment period, as assessed by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria through radiological imaging (CT/MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cao, MD, Principal Investigator — Division of Abdominal Tumor, Department of Medical Oncology, Cancer Center and State Key Laboratory of Biological Therapy, West China Hospital, Sichuan University, Chengdu, Sichuan
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy protection requirements, regulatory restrictions in China, and limitations in the original informed consent process that did not include provisions for external data sharing.